CLINICAL TRIAL: NCT04130971
Title: Predict - a Translational Study to Predict Tumour Response to Neoadjuvant Treatment
Brief Title: Predicting Colorectal Cancer - Tissue Samples to Evaluate Tumour Characteristics and Treatment Response
Acronym: Predict
Status: Recruiting | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Eva Angenete, PI, Sahlgrenska University Hospital
Other Study IDs: Predict
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Biopsies prior and after treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients without neoadjuvant treatment
  Interventions: Other: No intervention, just observation
- Patients with short course radiotherapy
  Interventions: Other: No intervention, just observation
- Patients with long course chemoradiotherapy
  Interventions: Other: No intervention, just observation
- Patients with short course radiotherapy and deferred surgery
  Interventions: Other: No intervention, just observation

INTERVENTIONS:
Other: No intervention, just observation — No intervention, just observation of the differences between groups and within patients.

SUMMARY:
All adult patients with colorectal cancer presenting within the Sahlgrenska University Hospital or treated at any time at Sahlgrenska University Hospital are eligible and will be asked to participate. We already have biopsies taken at surgery in patients that receive surgery, but this study will include all patients and the biopsies will be taken during endoscopy for diagnosis of the primary tumour. Biopsies will then be taken during follow-up exams prior surgery but after neoadjuvant treatment. Biopsies will also be taken during surgery and in cases where surgery is not necessary biopsies will be taken regularly during follow-up exams.

Blood samples and in relevant cases urinary samples and mouth swabs will be taken at all timepoints when biopsies are taken. If it is not possible to take biopsies prior treatment blood samples will still be drawn.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer

Exclusion Criteria:

* Not colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of colorectal cancer are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumour response to treatment | 1-2 months after initiated treatment
  Tumour microenviroment changes

SECONDARY OUTCOMES:
Normal tissue response to treatment | 1month -3 years after treatment
  Extra cellular matrix changes

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided